CLINICAL TRIAL: NCT04196621
Title: Clinical Evaluation of Reproducibility of Keratometric Measurements and Influencing Factors in Cataract Patients
Acronym: KerSty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2112/2018
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cataract; Dry Eye
MeSH Terms: conditions — Cataract; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Biometry will be performed in individuals with age related cataract. Patients will be classified as dry eye or normal eye. Two different artificial tears will be instilled at two time points in a randomized order with a time-lag of at least 24 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Which eye as well as the order of artificial eye drops will be randomized. Randomization information will be put in a sealed envelope on screening date and opened in operating theatre right before procedure start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High viscous artificial tears (Active Comparator): First, a native measurement at the IOL Master will be performed. Following which, high viscous artificial tears are installed and the biometry will be repeated within 30 seconds, as well as after 2 and 5 minutes
  Interventions: Device: High viscous artificial tears
- Low viscous artificial tears (Active Comparator): First, a native measurement at the IOL Master will be performed. Following which, low viscous artificial tears are installed and the biometry will be repeated within 30 seconds, as well as after 2 and 5 minutes
  Interventions: Device: Low viscous artificial tears

INTERVENTIONS:
Device: High viscous artificial tears — Instillation of one drop high viscous artificial tears
  Arms: High viscous artificial tears
Device: Low viscous artificial tears — Instillation of one drop low viscous artificial tears
  Arms: Low viscous artificial tears

SUMMARY:
The investigational device is an approved biometry device to perform biometric measurements preoperatively to calculate the needed IOL power.

First, two native measurements at the IOL Master will be performed. Thereafter randomly assigned artificial tears are instilled in the eye and biometry will be repeated within 30 seconds, as well as after 2 and 5 minutes.

At least 24hours after those measurements, two native measurements at the IOL Master will be performed. Thereafter, the not yet used artificial tears are instilled in the eye and biometry will be repeated within 30 seconds, as well as after 2 and 5 minutes.

Examinations will be implemented in accordance with the approved investigational plan on subjects and includes: repeated biometry without and with artificial tear drops.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed uni- or bilateral age-related cataract
* Age 40 to 95
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Corneal abnormality (Corneal scaring)
* usage of artificial tears/eyedrops 24h before the examination
* necessity of any topical therapy of the eye (i.e. glaucoma)
* active ocular or nasal allergies or corneal or conjunctival infection
* abnormality of the nasolacrimal drainage apparatus
* dry eye severity level 4 (severe and/or disabling constant discomfort and visual symptoms, marked conjunctival injection, filamentary keratitis, mucus clumping, tear debris, ulceration, trichiasis, keratinization, symblepharon)
* lid deformities
* Preceding ocular surgery or trauma
* Pregnancy
* Lactation
* Uncontrolled systemic or ocular disease

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine whether application of highly viscid eye drops in normal eyes leads to a change in keratometry measurements after 30 seconds. | 30 seconds
  The change in measured k-values (k, k1, k2 in mm) before and after instillation of artificial eye drops will be calculated

SECONDARY OUTCOMES:
To determine whether application of highly viscid eye drops in normal eyes leads to a change keratometry measurements after 2 minutes or 5 minutes. These objectives will be assessed analogously to the primary objective. | 2, 5minutes
  The change in measured k-values (k, k1, k2 in mm)before and after instillation of artificial eye drops will be calculated
To determine whether application of slightly viscid eye drops in normal and in dry eyes leads to a change in keratometry measurements after 30 seconds, 2 minutes or 5 minutes. These objectives will be assessed analogously to the primary objective | 30 seconds, 2 minutes or 5 minutes
  The change in measured k-values (k, k1, k2 in mm) before and after instillation of artificial eye drops will be calculated
To determine whether application of highly viscid eye drops in dry eyes leads to a change in keratometry measurements after 30 seconds, 2 minutes or 5 minutes. These objectives will be assessed analogously to the primary objective | 30 seconds, 2 minutes or 5 minutes
  The change in measured k-values (k, k1, k2 in mm) before and after instillation of artificial eye drops will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No